CLINICAL TRIAL: NCT04616209
Title: A Phase Ι & IIa, Open-label Study to Evaluate Safety and Efficacy of the Combination Therapy of Allogeneic PB103 and Standard Cancer Treatment in the IIIB/IV or Recurrent Non-small Cell Lung Cancer (NSCLC) Patients
Brief Title: Allogeneic PB103 (NK Cells) Therapy in Non-small Cell Lung Cancer (NSCLC) Patients
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Precision Biotech Taiwan Corp. (Industry)
Collaborators: Tri-Service General Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PB-2020Allo
Record Dates: First submitted 2020-10-08; First posted 2020-11-04 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Non-small Cell Lung Cancer
Keywords: allogeneic donor; NK cells
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PB103 (donor-derived NK cells) infusion (Experimental): Cohort 1: 0.5×10^9，Cohort 2:1×10^9 or Cohort 3: 1.5×10^9 cells
  Interventions: Biological: donor-derived NK cell infusion

INTERVENTIONS:
Biological: donor-derived NK cell infusion — PB103 administrations will be separated by 4-week interval

SUMMARY:
Objectives: To determine the safety, tolerability, and efficacy of allogeneic PB103 in patients with IIIb/IV or refractory non-small-cell lung cancer

DETAILED DESCRIPTION:
PB103 is allogeneic NK cells derived from a healthy donor. In this phase I/IIa trial, patients with IIIb/IV and refractory non-small cell lung cancer will be enrolled for testing the safety, tolerability, and efficacy of PB103 (NK cells). For assessment of safety and maximum tolerated dose (MTD) of PB103, three-dose levels of PB103 will be administered to enrolled patients based on the 3+3 dose-escalation design. MTD is deﬁned as one dose level below the dose at which dose-limiting toxicities (DLT) is observed in <33% of the participants. DLT is deﬁned as grade 4 toxicities (hematological toxicities), grade 3 toxicities (non-hematological toxicities), or acute GvHD more than grade 2. Once MTD is determined, 12 patients at MTD dose will be enrolled for assessment of safety and efficacy of PB103 at phase IIa.

ELIGIBILITY:
Inclusion Criteria:

Recipient:

1. Recipients (Subjects) are between 20-70 years of age.
2. Related donor: 6/6 matched at HLA-A, -B and -DRb1 or haploidentical donor ≥ 4/8 match at HLA-A, -B, -C and -DRb1
3. Signed informed consent.
4. Subjects with histologically or cytologically confirmed non -small-cell lung cancer of stage IIIB-IV, not amenable to definitive multi-modality therapy, or recurrent disease after a prior diagnosis of stage I-III disease. All staging is determined via the American Joint Committee on Cancer (AJCC)/IASLC 8th edition proposed staging criteria.
5. Subjects must have measurable or evaluable disease according to RECIST v1.1
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2.
7. Lifespan over 6 months.
8. Acceptable organ function, as evidenced by the following laboratory data:

（a） Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 3.0 × upper limit of normal (ULN). (for patients with known hepatic metastases, AST and/or ALT ≤ 5× ULN) （b） Total serum bilirubin ≤ 1.5 × ULN （c） Absolute neutrophil count (ANC) ≥ 1500 cells/mm3 （d） Platelet count ≥ 75,000 cells/mm3 （e） Hgb ≥ 9.0 g/dL （f） Estimated GFR ≥ 60 ml/min /1.73m2 or creatinine clearance ≥ 60 mL/min

Donor

1. Donors are between 20-65 years of age.
2. Related donor: 6/6 matched at HLA-A, -B and -DRb1 or haploidentical donor ≥ 4/8 match at HLA-A, -B, -C and -DRb1
3. Signed informed consent.

Exclusion Criteria:

Recipient:

1. Patients with history of clinically significant interstitial lung disease or radiation pneumonitis.
2. Patients with brain metastases or leptomeningeal disease.
3. Patients who have had radiation to the lung fields within four weeks of starting treatment. For all palliative radiation to all other sites, at least 7 days must have elapsed prior to starting to treatment.
4. Patients who have had major surgery (e.g., intra-thoracic, intra-abdominal, or intra-pelvic) within two weeks prior to starting study drug or who have not recovered from side effects of such procedure. Video-assisted thoracic surgery (VATS) and mediastinoscopy will not be counted as major surgery and patients can be enrolled in the study ≥1 week after the procedure.
5. Patients who received anti-cancer treatment and did not recover from toxicities to grades 0-1 by NCI CTCAE (version 5.0) are not eligible but WBC and Hgb Grade 2 is acceptable.
6. Patients with a second, clinically active, cancer. Patients with second cancers that have been treated with curative intent and/or are currently inactive are allowed.
7. Known history of human immunodeficiency virus (HIV) seropositivity.
8. Participants who are receiving any other investigational agents. Patients previously treated with investigational agents must complete a washout period of at least one week or five half-lives, whichever is longer, before starting treatment.
9. Patients receiving concomitant immunosuppressive agents or chronic corticosteroid use, except those on topical or inhaled steroids, or steroids are given via local injection.
10. Patients with clinically significant, uncontrolled cardiovascular disease, such as unstable angina or myocardial infarction within 6 months prior to screening, abnormal left ventricular ejection fraction (LVEF <50%), cardiac arrhythmia not controlled with medication, uncontrolled hypertension defined as an SBP ≥ 160mm Hg and/or DBP ≥ 100mm Hg, with or without anti-hypertensive medication. Initiation or adjustment of antihypertensive medication(s) is allowed prior to screening.
11. Presence of fungal, bacterial, viral, or other infection requiring IV antimicrobials for management.
12. Pregnancy and lactating women.
13. Other situations the investigators think not eligible for participation in the research.

Donor

1. Donors who are pregnant and lactating women.
2. Donor who has had advanced tumor diseases.
3. Donor who has had autoimmune diseases.
4. Donors are positive for one of human immunodeficiency virus (HIV), syphilis serology test (RPR+TPHA), CMV IgM, human T-lymphotropic virus (HTLV), and hepatitis B and C virus.
5. Other situations the investigators think not eligible for participation in the research.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2020-11-15 (Actual); Primary Completion 2027-12-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
safety of PB103 | one year
  assessment of adverse events

SECONDARY OUTCOMES:
efficacy of PB103 | one year
  assessment of Progression Free Survival, PFS

CONTACTS AND LOCATIONS:
Overall Officials: Ming-Shen Dai, MD/PhD, Principal Investigator — Tri-Service General Hospital
Locations (1):
- Tri-Service General Hospital, Taipei, Taiwan